CLINICAL TRIAL: NCT04736602
Title: An Open-label, Multicentre, Single Arm Study to Assess the Efficacy and Safety of Triptorelin 3-month Formulation in Chinese Children With Central Precocious Puberty
Brief Title: Efficacy and Safety Study of Triptorelin 3-Month Formulation in Chinese Children With Central Precocious Puberty.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-CN-52014-243
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triptorelin Pamoate 15mg for injection (Experimental): Triptorelin was injected at day 1 and month 3.
  If participants were willing to enter the extension phase, two additional Triptorelin injections were given at month 6 and month 9.
  Interventions: Drug: Triptorelin pamoate 15mg

INTERVENTIONS:
Drug: Triptorelin pamoate 15mg — Intramuscular injection (IM)

SUMMARY:
The purpose of this research was to confirm the effectiveness and safety of the study drug, Triptorelin pamoate 15mg 3-month formulation, in a Chinese population of Central Precocious Puberty (CPP) children.

ELIGIBILITY:
Inclusion Criteria:

* Onset of development of secondary sex characteristics before 8 and 9 years in girls and boys, respectively breast development in girls or testicular enlargement in boys according to the Tanner method: Stage II
* Pubertal response of LH to GnRH stimulation test (stimulated peak LH ≥5 IU/L)
* Difference between bone age (BA) (according to Greulich and Pyle method) and chronological age (CA) >1 year
* Girls with Tanner staging ≥2 for breast development and enlarged uterine length and several follicles with diameter >4 mm in the ovary at Screening visit; boys who have testicular volume ≥4 mL at Screening visit
* Age < 9 years old for girls and < 10 years old for boys at initiation of triptorelin treatment
* Weight at least 20 kg
* Subjects will qualify for the extension phase if they sign the corresponding specific consent form, are still benefiting from treatment at the end the primary study and have not experienced any unacceptable safety issues.

Exclusion Criteria:

* Gonadotropin-independent (peripheral) precocious puberty: extra pituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroid secretion
* Non-progressing isolated premature thelarche
* Presence of an unstable intracranial tumour or an intracranial tumour requiring neurosurgery or cerebral irradiation. Participants with hamartomas not requiring surgery are eligible
* Evidence of renal (creatinine >1.5 x upper limit of normal (ULN)) or hepatic impairment (bilirubin >1.5 x ULN or alanine aminotransferase (ALT)/aspartate transaminase (AST) >3 x ULN)
* Any other condition or chronic illness or treatment possibly interfering with growth or other study endpoints (e.g. chronic steroid use except topical steroids, renal failure, diabetes, moderate to severe scoliosis)
* Prior or current therapy with a GnRH agonist (GnRHa), medroxyprogesterone acetate, growth hormone or insulin-like growth factor-1 (IGF-1)
* Diagnosis of short stature, i.e. >2.25 standard deviation (SD) below the mean height for age
* Major medical or psychiatric illness that could interfere with study visits
* Known hypersensitivity to any of the test materials or related compounds
* Use of anticoagulants (heparin and coumarin derivatives) within the 2 weeks prior to the Screening visit.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- China (7):
  - Chengdu Women's and Children's Central Hospital, Chengdu
  - Jiangxi Provincial Children's Hospital, Nanchang
  - Children's Hospital of Nanjing, Nanjing
  - Tangshan Maternal & Child Health Hospital, Tangshan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan
  - Wuxi Children's Hospital, Wuxi
  - Henan Children's Hospital, Zhengzhou Children's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, Phase 3, open-label, single arm, 2-phase (main study phase and an extension phase) study was conducted in children with central precocious puberty (CPP) at 6 investigational sites in China.
Pre-assignment Details: This study consisted of screening period (up to 28 days), main study phase (6 months) and an optional extension phase (6 months). A total of 32 participants were enrolled in this study.
Groups:
- All Participants: Participants received triptorelin pamoate 15 milligrams (mg) intramuscular (IM) injection on Day 1 visit and Month 3 visit (Day 91) during the main study phase. Participants had an option to continue with the triptorelin pamoate in extension phase of the study. As per Investigator decision, eligible participants continued to receive IM injections of triptorelin pamoate on Month 6 (Day 182) and Month 9 (Day 271) during the extension phase.
Period: Main Study Phase
Arm/Group | All Participants
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Parent/Guardian | 2
Period: Extension Phase
Arm/Group | All Participants
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Parent/Guardian | 1

BASELINE CHARACTERISTICS:
Population: Intention-To-Treat (ITT) population consisted of all participants who received at least 1 dose of study medication.
Groups:
- All Participants: Participants received triptorelin pamoate 15 mg IM injection on Day 1 visit and Month 3 visit (Day 91) during the main study phase. Participants had an option to continue with the triptorelin pamoate in extension phase of the study. As per Investigator decision, eligible participants continued to receive IM injections of triptorelin pamoate on Month 6 (Day 182) and Month 9 (Day 271) during the extension phase.
Arm/Group | All Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Luteinising Hormone (LH) Suppression After Gonadotropin-Releasing Hormone (GnRH) Stimulation
Description: The LH suppression was defined as stimulated peak LH ≤3 International Units/Liter (IU/L). The GnRH stimulation test was performed by using an intravenous (IV) injection of gonadorelin (synthetic GnRH) to stimulate gonadotrophin release and blood samples were collected after the gonadorelin injection for central assessment of serum LH levels.
Time Frame: At Month 3
Population: The modified ITT (mITT) population consisted of all treated participants with at least 1 baseline and Month 3 post-baseline assessment of the primary efficacy endpoint.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants | 100 [90.8 to 100]

2. Secondary Outcome: Change From Baseline in Basal LH and Follicle-Stimulating Hormone (FSH) Serum Levels
Description: Basal LH and FSH serum concentrations were analyzed centrally. Change from baseline was defined as the value for LH and FSH levels at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6, 9 and 12
Population: The mITT population consisted of all treated participants with at least 1 baseline and Month 3 post-baseline assessment of the primary efficacy endpoint. Only data from the participants analyzed were reported.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | All Participants
Number analyzed (Participants) | 31
IU/L
  LH, Month 3 | -0.6906 (1.6417)
  LH, Month 6: number analyzed (Participants) | 30
  LH, Month 6 | -0.7411 (1.6606)
  LH, Month 9: number analyzed (Participants) | 28
  LH, Month 9 | -0.7415 (1.6817)
  LH, Month 12: number analyzed (Participants) | 29
  LH, Month 12 | -0.9310 (1.6367)
  FSH, Month 3 | -2.3531 (1.8079)
  FSH, Month 6: number analyzed (Participants) | 30
  FSH, Month 6 | -2.2307 (1.7445)
  FSH, Month 9: number analyzed (Participants) | 28
  FSH, Month 9 | -2.0740 (1.7979)
  FSH, Month 12: number analyzed (Participants) | 29
  FSH, Month 12 | -1.9413 (1.6996)

3. Secondary Outcome: Percentage of Participants With LH Suppression After GnRH Stimulation
Description: A synthetic GnRH (gonadorelin) was used for gonadotrophin stimulation. Blood samples were collected prior to gonadorelin injection (timepoint T0) and at 30 minutes (T30), 60 minutes (T60) and 90 minutes (T90) (±5 minutes at each timepoint) after a single IV injection of gonadorelin. A suppressed LH response to GnRH stimulation test was defined as peak LH ≤3 IU/L among the 4 timepoints T0, T30, T60 and T90).
Time Frame: At Months 6 and 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
percentage of participants
  Month 6 | 93.5 [81.1 to 98.8]
  Month 12 | 93.5 [81.1 to 98.8]

4. Secondary Outcome: Change From Baseline in Peak LH and FSH Level After GnRH Stimulation
Description: A synthetic GnRH was used for gonadotrophin stimulation. Blood samples were collected prior to gonadorelin injection (timepoint T0) and at 30 minutes (T30), 60 minutes (T60) and 90 minutes (T90) (±5 minutes at each timepoint) after a single IV injection of gonadorelin. The FSH response to GnRH stimulation was the peak FSH level among the 4 timepoints (T0, T30, T60 and T90). The LH response to GnRH stimulation test was defined as peak LH ≤3 IU/L among the 4 timepoints T0, T30, T60 and T90). Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | All Participants
Number analyzed (Participants) | 31
IU/L
  LH, Month 3 | -23.0969 (17.9856)
  LH, Month 6: number analyzed (Participants) | 29
  LH, Month 6 | -24.3596 (17.9180)
  LH, Month 12: number analyzed (Participants) | 29
  LH, Month 12 | -23.7221 (18.3669)
  FSH, Month 3 | -11.2757 (4.5026)
  FSH, Month 6: number analyzed (Participants) | 29
  FSH, Month 6 | -11.2536 (4.5267)
  FSH, Month 12: number analyzed (Participants) | 29
  FSH, Month 12 | -10.4701 (4.8424)

5. Secondary Outcome: Percentage of Participants With Prepubertal Levels of Sex Steroids
Description: Prepubertal sex steroids assessment included estradiol in female participants and testosterone in male participants. Prepubertal sex steroids levels were defined as: estradiol ≤20 picogram (pg)/milliliter (mL) in female participants and testosterone ≤0.3 nanogram (ng)/mL in male participants.
Time Frame: At Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants
  Month 3 | 100 [90.8 to 100]
  Month 6: number analyzed (Participants) | 30
  Month 6 | 96.8 [85.6 to 99.8]
  Month 9: number analyzed (Participants) | 28
  Month 9 | 90.3 [76.8 to 97.3]
  Month 12: number analyzed (Participants) | 29
  Month 12 | 93.5 [81.1 to 98.8]

6. Secondary Outcome: Change From Baseline in Estradiol Levels
Description: Estradiol serum concentration was analyzed centrally. Change from baseline was defined as the value for estradiol levels at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6 ,9 and 12
Population: The mITT population consisted of all treated participants with at least 1 baseline and Month 3 post-baseline assessment of the primary efficacy endpoint. Only data for female participants were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 28
pg/mL
  Month 3 | -8.0047 (15.6905)
  Month 6: number analyzed (Participants) | 27
  Month 6 | -8.3011 (15.9093)
  Month 9: number analyzed (Participants) | 25
  Month 9 | -7.7458 (15.8683)
  Month 12: number analyzed (Participants) | 26
  Month 12 | -8.6204 (16.1359)

7. Secondary Outcome: Change From Baseline in Testosterone Levels
Description: Testosterone serum concentration was analyzed centrally. Change from baseline was defined as the value for testosterone levels at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6 ,9 and 12
Population: The mITT population consisted of all treated participants with at least 1 baseline and Month 3 post-baseline assessment of the primary efficacy endpoint. Only data for male participants were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All Participants
Number analyzed (Participants) | 3
ng/mL
  Month 3 | -1.3650 (1.1734)
  Month 6 | -1.3650 (1.1734)
  Month 9 | -1.3650 (1.1734)
  Month 12 | -1.3650 (1.1734)

8. Secondary Outcome: Percentage of Participants With Change From Baseline in Pubertal Stage
Description: Pubertal stage parameters were analyzed using Tanner method. Pubertal stage parameters included genital stage in male participants, breast stage in female participants and pubic hair stage in both sexes.
Time Frame: Baseline (Day 1) and at Months 6 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants
  Breast development stage for female participants, Month 6, No change: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 6, No change | 35.7
  Breast development stage for female participants, Month 6, Reduced: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 6, Reduced | 57.1
  Breast development stage for female participants, Month 6, Increased: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 6, Increased | 3.6
  Breast development stage for female participants, Month 6, Missing: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 6, Missing | 3.6
  Genital development stage for male participants, Month 6, No change: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 6, No change | 33.3
  Genital development stage for male participants, Month 6, Reduced: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 6, Reduced | 66.7
  Genital development stage for male participants, Month 6, Increased: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 6, Increased | 0
  Genital development stage for male participants, Month 6, Missing: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 6, Missing | 0
  Pubic hair development stage for female participants, Month 6, No change: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 6, No change | 96.4
  Pubic hair development stage for female participants, Month 6, Reduced: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 6, Reduced | 0
  Pubic hair development stage for female participants, Month 6, Increased: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 6, Increased | 0
  Pubic hair development stage for female participants, Month 6, Missing: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 6, Missing | 3.6
  Pubic hair development stage for male participants, Month 6, No change: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 6, No change | 66.7
  Pubic hair development stage for male participants, Month 6, Reduced: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 6, Reduced | 33.3
  Pubic hair development stage for male participants, Month 6, Increased: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 6, Increased | 0
  Pubic hair development stage for male participants, Month 6, Missing: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 6, Missing | 0
  Breast development stage for female participants, Month 12, No change: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 12, No change | 39.3
  Breast development stage for female participants, Month 12, Reduced: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 12, Reduced | 50.0
  Breast development stage for female participants, Month 12, Increased: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 12, Increased | 3.6
  Breast development stage for female participants, Month 12, Missing: number analyzed (Participants) | 28
  Breast development stage for female participants, Month 12, Missing | 7.1
  Genital development stage for male participants, Month 12, No change: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 12, No change | 0
  Genital development stage for male participants, Month 12, Reduced: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 12, Reduced | 100
  Genital development stage for male participants, Month 12, Increased: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 12, Increased | 0
  Genital development stage for male participants, Month 12, Missing: number analyzed (Participants) | 3
  Genital development stage for male participants, Month 12, Missing | 0
  Pubic hair development stage for female participants, Month 12, No change: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 12, No change | 82.1
  Pubic hair development stage for female participants, Month 12, Reduced: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 12, Reduced | 0
  Pubic hair development stage for female participants, Month 12, Increased: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 12, Increased | 10.7
  Pubic hair development stage for female participants, Month 12, Missing: number analyzed (Participants) | 28
  Pubic hair development stage for female participants, Month 12, Missing | 7.1
  Pubic hair development stage for male participants, Month 12, No change: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 12, No change | 66.7
  Pubic hair development stage for male participants, Month 12, Reduced: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 12, Reduced | 33.3
  Pubic hair development stage for male participants, Month 12, Increased: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 12, Increased | 0
  Pubic hair development stage for male participants, Month 12, Missing: number analyzed (Participants) | 3
  Pubic hair development stage for male participants, Month 12, Missing | 0

9. Secondary Outcome: Percentage of Participants With Stabilized Pubertal Stage Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline (Day 1) and at Months 6 and 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants
  Breast development stage for girls, Month 6: number analyzed (Participants) | 27
  Breast development stage for girls, Month 6 | 92.9 [79.2 to 98.7]
  Genital development stage for boys, Month 6: number analyzed (Participants) | 3
  Genital development stage for boys, Month 6 | 100 [36.8 to 100.0]
  Pubic hair development stage for girls, Month 6: number analyzed (Participants) | 27
  Pubic hair development stage for girls, Month 6 | 96.4 [84.1 to 99.8]
  Pubic hair development stage for boys, Month 6: number analyzed (Participants) | 3
  Pubic hair development stage for boys, Month 6 | 100 [36.8 to 100.0]
  Breast development stage for girls, Month 12: number analyzed (Participants) | 26
  Breast development stage for girls, Month 12 | 89.3 [74.6 to 97.0]
  Genital development stage for boys, Month 12: number analyzed (Participants) | 3
  Genital development stage for boys, Month 12 | 100 [36.8 to 100.0]
  Pubic hair development stage for girls, Month 12: number analyzed (Participants) | 26
  Pubic hair development stage for girls, Month 12 | 82.1 [66.1 to 92.7]
  Pubic hair development stage for boys, Month 12: number analyzed (Participants) | 3
  Pubic hair development stage for boys, Month 12 | 100 [36.8 to 100.0]

10. Secondary Outcome: Change From Baseline in Auxological Parameter: Height
Description: Auxological parameter including height was analyzed. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | All Participants
Number analyzed (Participants) | 31
centimeter (cm)
  Month 3 | 2.24 (0.62)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 3.55 (0.69)
  Month 9: number analyzed (Participants) | 30
  Month 9 | 4.63 (0.81)
  Month 12: number analyzed (Participants) | 29
  Month 12 | 6.54 (0.88)

11. Secondary Outcome: Change From Baseline in Auxological Parameter: Weight
Description: Auxological parameter including weight was analyzed. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | All Participants
Number analyzed (Participants) | 31
kilogram (kg)
  Month 3 | 1.284 (1.319)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 2.533 (1.647)
  Month 9: number analyzed (Participants) | 30
  Month 9 | 3.290 (1.899)
  Month 12: number analyzed (Participants) | 29
  Month 12 | 4.818 (2.385)

12. Secondary Outcome: Change From Baseline in Auxological Parameter: Growth Velocity
Description: Auxological parameter including growth velocity was analyzed. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | All Participants
Number analyzed (Participants) | 31
cm/year
  Month 3 | -0.895 (3.637)
  Month 6: number analyzed (Participants) | 30
  Month 6 | -3.769 (2.806)
  Month 9: number analyzed (Participants) | 30
  Month 9 | -4.804 (2.927)
  Month 12: number analyzed (Participants) | 29
  Month 12 | -2.052 (3.089)

13. Secondary Outcome: Change From Baseline in Auxological Parameter: Body Mass Index (BMI)
Description: Auxological parameter including BMI was analyzed. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/meter square
Arm/Group | All Participants
Number analyzed (Participants) | 31
kg/meter square
  Month 3 | 0.142 (0.702)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 0.470 (0.791)
  Month 9: number analyzed (Participants) | 30
  Month 9 | 0.585 (0.849)
  Month 12: number analyzed (Participants) | 29
  Month 12 | 0.895 (1.081)

14. Secondary Outcome: Change From Baseline in Bone Age (BA)
Description: BA was determined using X-rays of the hand and wrist. Change from baseline was defined as the value for BA at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 30
years
  Month 6 | 0.233 (0.307)
  Month 12: number analyzed (Participants) | 29
  Month 12 | 0.586 (0.544)

15. Secondary Outcome: Change From Baseline Difference Between BA and Chronological Age (CA)
Description: BA was determined using X-rays of the hand and wrist. Change from baseline was defined as the difference between BA and CA value at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 30
years
  Month 6 | -0.44 (0.53)
  Month 12: number analyzed (Participants) | 29
  Month 12 | -0.48 (0.57)

16. Secondary Outcome: Change From Baseline in Uterine Length
Description: Uterine length was determined by type B ultrasound. Change from baseline was defined as the value of uterine length at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 6 and12
Population: The mITT population consisted of all treated participants with at least 1 baseline and Month 3 post-baseline assessment of the primary efficacy endpoint. Only data from the female participants analyzed were reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 28
cm
  Month 6: number analyzed (Participants) | 26
  Month 6 | -0.4012 (0.4391)
  Month 12: number analyzed (Participants) | 24
  Month 12 | -0.3771 (0.6534)

17. Secondary Outcome: Change From Baseline of Testicular Volume
Description: Testicular volume was determined by type B ultrasound. Change from baseline was defined as the value of testicular volume at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first dose administered.
Time Frame: Baseline (Day 1) and at Months 6 and 12
Population: The mITT population consisted of all treated participants with at least 1 baseline and Month 3 post-baseline assessment of the primary efficacy endpoint. Only data from the male participants analyzed were reported. The Number Analyzed for left and right are not consistent for each month because one participant did not have the examination on the left testicular throughout the study.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | All Participants
Number analyzed (Participants) | 3
mL
  Left, Month 6: number analyzed (Participants) | 2
  Left, Month 6 | -2.4022 (1.7109)
  Right, Month 6 | -4.7334 (4.4222)
  Left, Month 12: number analyzed (Participants) | 1
  Left, Month 12 | -2.8840 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed.
  Right, Month 12: number analyzed (Participants) | 2
  Right, Month 12 | -6.7975 (6.3958)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported from the first dose of study treatment (Day 1) up to end of extension phase, a maximum of approximately 368 days.
Description: Safety population consisted of all participants who received at least 1 dose of study medication and had at least 1 post-baseline safety assessment.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=32)
Pneumonia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=32)
Upper respiratory tract infection (Infections and infestations) | 10 (15)
Bronchitis (Infections and infestations) | 3 (4)
Tonsillitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 7 (7)
Overweight (Metabolism and nutrition disorders) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 2 (2)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Retained deciduous tooth (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Chest discomfort (General disorders) | 1 (2)
Condition aggravated (General disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Red blood cells urine (Investigations) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tic (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT04736602/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT04736602/SAP_001.pdf